CLINICAL TRIAL: NCT07071272
Title: Non-inferiority Study of Mammography With the Contrast Medium (Contrast-enhanced Digital Mammography, CEDM) Versus Breast Magnetic Resonance (MRI)
Brief Title: Non-inferiority Study of Contrast-enhanced Digital Mammography (CEDM) vs Magnetic Resonance Imaging (MRI) in Terms of Diagnostic Accuracy in Patients Undergoing Preoperative Staging of Established Invasive Breast Cancer
Acronym: CEDM-VR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CEDM-VR-2803CESC
Record Dates: First submitted 2025-05-13; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: CEM; breast cancer; breast MR
MeSH Terms: conditions — Breast Neoplasms | interventions — omega-Chloroacetophenone

STUDY DESIGN:
Intervention Model Description: Participants will undergo a routine clinical MRI followed by CEDM during a scheduled visit. Imaging will be interpreted independently by two radiologists, blinded to each other's findings, with subsequent consensus reporting. Pseudonymized data will be recorded, including imaging findings, histological results, and any adverse reactions to contrast agents.
  In group 2 (neoadjuvant chemotherapy), patients will also undergo interim imaging with both MRI and CEDM at 3 and 6 months to assess treatment response.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing preoperative staging and patients undergoing chemotherapy (Experimental): All participants in the group 1 and 2 will undergo a routine clinical MRI followed by CEM during a scheduled visit.
  In group 2 (neoadjuvant chemotherapy), patients will also undergo interim imaging with both MRI and CEDM at 3 and 6 months to assess treatment response.
  Interventions: Other: breast-MRI and CEM

INTERVENTIONS:
Other: breast-MRI and CEM — Participants will undergo a breast MRI followed by CEM for local breast cancer staging

SUMMARY:
The general objective of the study is to verify the diagnostic accuracy of contrast-enhanced mammography (CEM) compared to breast magnetic resonance imaging in patients undergoing preoperative staging for breast neoformations that have already been diagnosed and in patients undergoing neoadjuvant chemotherapy.

In addition to performing a preoperative breast resonance imaging, which is always performed in these patients, one contrast-enhanced mammography per patient is planned.

In patients undergoing neoadjuvant chemotherapy, which usually undergo MRI examination at the beginning, mid-cycle and at the end of chemotherapy treatment, a CEM will also be acquired same way at the beginning, mid-cycle and at the end of chemotherapy treatment.

The study requires, for the execution of the contrast-enhanced mammography exam, the administration of an iodinated contrast medium that is completely analogous to that used in computed tomography.

DETAILED DESCRIPTION:
This is a monocentric, prospective, experimental non-inferiority study evaluating the diagnostic performance of Contrast-Enhanced Digital Mammography (CEDM/CEM) compared to Breast Magnetic Resonance Imaging (MRI) in the preoperative assessment and staging of breast cancer.

MRI, recognized for its high sensitivity and three-dimensional visualization capabilities without ionizing radiation, is often used in specialized centers for detailed staging. However, it suffers from practical limitations including high cost, long exam duration (~7-10 minutes), and cost-effective. Preliminary studies suggest its diagnostic accuracy may be comparable to, or even better than, MRI, especially regarding specificity and lesion size estimation. Furthermore, CEM can be used in patients with contraindications to MRI, including those with pacemakers, cochlear implants, or severe claustrophobia.

The study will enroll approximately 216 patients up to December 2025, divided in tho groups: 108 patients with already confirmed invasive breast cancer undergoing preoperative staging; 108 patients scheduled for neoadjuvant chemotherapy followed by surgery.

CEM and MRI will be performed for all enrolled participants. Histological examination of biopsy or surgical specimens will serve as the reference standard for evaluating diagnostic performance.

The primary outcome is to determine diagnostic accuracy (including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV)) of CEDM versus MRI, using histopathology as the gold standard. A non-inferiority margin (Δ) of 15% is defined. The non-inferiority hypothesis will be tested using paired binary outcomes, and sample size calculations for groups 1 and 2, accounting for dependent diagnostic testing.

The secondary endpoint are:

* evaluating interobserver agreement between radiologists interpreting CEDM (Cohen's kappa and intraclass correlation coefficients).
* comparison of lesion size estimations and regression evaluations in patients undergoing neoadjuvant chemotherapy at baseline (T0), 3 months (T3), and 6 months (T6).

Descriptive statistics will summarize demographic and clinical characteristics. For hypothesis testing, paired comparisons will be used: Student's t-test or Wilcoxon test for continuous variables; McNemar test or Fisher's exact test for categorical variables. Pearson correlation coefficients will assess the relationship between imaging measurements and histology. Diagnostic accuracy comparisons will assess the lower bound of the 95% confidence interval against the non-inferiority threshold.

Participants must be women over 30 years of age with a BI-RADS mammographic pattern >1, scheduled for a diagnostic MRI and meeting one of the five group classifications. Key exclusion criteria include: breast implants, known BRCA1 or BRCA2 mutations, contraindications to MRI, or impaired renal function (eGFR <30 mL/min). All participants must provide informed consent.

Participants will undergo a routine clinical MRI followed by CEDM during a scheduled visit. Imaging will be interpreted independently by two radiologists, blinded to each other's findings, with subsequent consensus reporting. Pseudonymized data will be recorded, including imaging findings, histological results, and any adverse reactions to contrast agents.

In group 2 (neoadjuvant chemotherapy), patients will also undergo interim imaging with both MRI and CEDM at 3 and 6 months to assess treatment response.

ELIGIBILITY:
Inclusion Criteria:

* women in pre-hospitalization with already established invasive breast cancer (T1-2)
* over the age of 30
* with BI-RADS mammography pattern> 1
* Written and signed informed consent for research
* Negative history of adverse events to the use of iodinated and chelated contrast media of gadolinium
* No significant renal impairment (EGFR> 30 mL / min within three months before administration of the iodinated contrast medium)

Exclusion Criteria:

* women with breast implants
* women under the age of 30
* Any contraindication to performing the MRI exam
* Women with known BRCA 1 and BRCA 2 mutation

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of the CEDM against breast MRI | Time Frame: Up to 6 months from baseline imaging (MRI and CEDM)
  The primary outcome is to assess diagnostic accuracy (including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV)) of CEDM versus MRI, using histopathology as the gold standard. A non-inferiority margin (Δ) of 15% is defined. The non-inferiority hypothesis will be tested using paired binary outcomes, and sample size calculations for groups 1 and 2 follow the Liu et al. method, accounting for dependent diagnostic testing.

SECONDARY OUTCOMES:
Inter-observer agreement | At baseline imaging (single time point)
  Assessment of interobserver agreement between radiologists interpreting CEDM using Cohen's kappa for categorical assessments and ICC for continuous variables (e.g., lesion size).
  Unit of Measure: Agreement coefficients (kappa, ICC)
Tumor size and regression evaluation (neoadjuvant patients) | Up to 6 months per participant
  Comparison of lesion size estimation and tumor regression in neoadjuvant chemotherapy patients at baseline (T0), 3 months (T3), and 6 months (T6).
  Unit of Measure: Lesion size in millimeters (mm); tumor regression in percentage (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Borgo Trento, AOUI Verona, Verona, Italy, Italy